CLINICAL TRIAL: NCT06785558
Title: The Role of Urinary ATP in the Diagnosis, Treatment, and Follow-up of Children with Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MAR.UAD.0012
Record Dates: First submitted 2024-12-23; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Overactive Bladder (OAB)
Keywords: Overactive bladder, urinary ATP, pediatric urology
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Control Group (No Intervention): The study include healthy control group with 10 child who haven't overactive bladder symptoms
- Overactive Bladder Group (Active Comparator): 30 child wit overactive bladder symptoms
  Interventions: Drug: Anticholinergic therapy

INTERVENTIONS:
Drug: Anticholinergic therapy — Overactive bladder group use anticholinergic drug and 1 month later their urinary atp levels calculated again
  Arms: Overactive Bladder Group

SUMMARY:
In this study, the investigators aim to evaluate the role of urinary ATP as a biomarker for the diagnosis, treatment, and follow-up of OAB in children for the first time in a clinical investigation, as previous research has been limited to adults.

DETAILED DESCRIPTION:
The diagnosis of OAB primarily relies on **medical history** and **physical examination**. Diagnosis is supported by appropriate laboratory findings and imaging methods. The role of various urinary biomarkers has been investigated as a non-invasive and simple diagnostic method. In recent years, research has focused on several biomarkers, particularly low-grade inflammatory mediators such as cytokines, Prostaglandin E2 (PGE2), Nerve Growth Factor (NGF), and Brain-Derived Neurotrophic Factor (BDNF). However, although these biomarkers are correlated with the severity of OAB symptoms, no studies have demonstrated their independent prognostic value.

For example, some studies report significant variability in urinary NGF levels, with not all patients showing increased urinary NGF. Other studies have noted that NGF correlates with OAB symptoms and decreases significantly after treatment. Consequently, no biomarker has yet been defined for routine clinical use. Moreover, biomarker studies specifically targeting pediatric OAB are limited, with most research focusing on adult populations and extrapolating findings to children.

Today, there is growing recognition of the role of purinergic transmission in urinary dysfunction. Purinergic transmission involves both afferent and efferent pathways in bladder emptying and has been implicated in the pathogenesis of detrusor overactivity (DO). In vitro studies have demonstrated that bladders with DO release higher amounts of Adenosine Triphosphate (ATP) from urothelium and cholinergic nerve terminals compared to normal bladders. Clinical studies suggest that urinary ATP levels could serve as a potential biomarker for OAB in adults. However, our literature review revealed that this biomarker has not yet been evaluated in children with OAB.

In this study, the investigators aim to evaluate the role of urinary ATP as a biomarker for the diagnosis, treatment, and follow-up of OAB in children for the first time in a clinical investigation, as previous research has been limited to adults.

Two midstream urine samples will collected from the OAB group: one pre-treatment and one at the first month of anticholinergic treatment. Urine samples will centrifuged, stored at -80°C, and ATP levels will measure via ELISA. Comparisons will make between the groups and pre-/post-treatment ATP levels in the OAB group. Correlation analysis will conduct between ATP levels and lower urinary system (LUS) parameters.

ELIGIBILITY:
Inclusion Criteria:

* The patient is under 18 years of age
* OAB symptoms may be accompanied by frequent urination, urgency, and urinary incontinence

Exclusion Criteria:

* Neurological disease
* malignancy
* active urinary tract infection
* bladder anomaly (uroterocele, diverticulum),
* LUS obstruction, ectopic ureter
* history of previous urological surgery

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Urinary ATP levels | Baseline

SECONDARY OUTCOMES:
Urinary ATP levels | 1 month
  Measured only overactive bladder group

CONTACTS AND LOCATIONS:
Overall Officials: CAGRI AKIN SEKERCİ, Study Director — MARMARA UNİVERSİTY SCHOOL OF MEDİCİNE DEPARTMENT OF UROLOGY
Locations (1):
- Marmara University School of Medicine Urology Department, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seltzsam S, Wang C, Zheng B, Mann N, Connaughton DM, Wu CW, Schneider S, Schierbaum L, Kause F, Kolvenbach CM, Nakayama M, Dai R, Ottlewski I, Schneider R, Deutsch K, Buerger F, Klambt V, Mao Y, Onuchic-Whitford AC, Nicolas-Frank C, Yousef K, Pantel D, Lai EW, Salmanullah D, Majmundar AJ, Bauer SB, Rodig NM, Somers MJG, Traum AZ, Stein DR, Daga A, Baum MA, Daouk GH, Tasic V, Awad HS, Eid LA, El Desoky S, Shalaby M, Kari JA, Fathy HM, Soliman NA, Mane SM, Shril S, Ferguson MA, Hildebrandt F. Reverse phenotyping facilitates disease allele calling in exome sequencing of patients with CAKUT. Genet Med. 2022 Feb;24(2):307-318. doi: 10.1016/j.gim.2021.09.010. Epub 2021 Nov 30. PMID 34906515
- [Derived] Altuntas T, Sekerci CA, Basok BI, Fidan M, Ozkan OC, Yucel S, Cam K, Tarcan T. The Role of Urinary ATP in the Diagnosis, Treatment, and Follow-up of Children With Overactive Bladder. Neurourol Urodyn. 2026 Jan;45(1):218-224. doi: 10.1002/nau.70168. Epub 2025 Oct 15. PMID 41097836